CLINICAL TRIAL: NCT02575651
Title: A Phase I, Open-label, Dose Escalation Study to Assess the Safety and Tolerability of Fluzoparib Following Single and Multiple Oral Doses in Patients With Advanced Solid Malignancies
Brief Title: A Phase I Study of Fluzoparib in Patient With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: 307 Hospital of PLA (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-FZPL-I-AST-TOL/PK
Record Dates: First submitted 2015-10-08; First posted 2015-10-15 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Advanced Solid Malignancies
Keywords: PARP; Advanced Solid Malignancies; Fluzoparib; Ovarian Cancer; BRCA
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluzoparib (Experimental): Each subject will receive a single dose of fluzoparib on day 1, and then subject will receive fluzoparib twice daily for 28 days during cycle 1.
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib either at 10,20,40,80,120mg ....., capsule oral.

SUMMARY:
Fluzoparib is an oral potent, selective PARP-1 and PARP-2 inhibitor. The objective of this study will be to investigate the safety and tolerability of Fluzoparib Capsule when given orally to Chinese patients with advanced solid malignancies. In addition, the pharmacokinetic profile, MTD (if possible) and efficacy of Fluzoparib will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 to 1.
* Life expectancy of more than 12 weeks.
* At least one measurable lesion exists.(RECIST 1.1).
* Subjects diagnosed with advanced solid malignancies who are refractory to standard therapies or for which no standard therapy exists.
* Subjects who have overall good overall general condition.
* Signed informed consent.

Exclusion Criteria:

* Subjects who received any previous treatment with a PARP inhibitor.
* Less than 4 weeks from the last clinical trial.
* Less than 4 weeks from the last radiotherapy, chemotherapy, surgery, hermone treatment and target therapy.
* Subjects that are unable to swallow, or dysfunction of gastrointestinal absorption.
* Subjects with symptomatic uncontrolled brain metastases.
* Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry.
* Subjects with a known hypersensitivity to Fluzoparib or any of the excipients of the product.
* Ongoing infection (determined by investigator).
* History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation.
* Subjects who can not interrupt the using of the drugs that may cause QT prolongation during study.
* Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial.
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The maximum-tolerated dose (MTD) will be defined as the maximum dose level at which no more than one subject out of three experiences has a dose-limiting toxicity (DLT) upon completing one treatment cycle. | 4 weeks

SECONDARY OUTCOMES:
Evaluation of pharmacokinetic parameter of Fluzoparib: Cmax | 4 weeks
Evaluation of pharmacokinetic parameter of Fluzoparib: Tmax | 4 weeks
Evaluation of pharmacokinetic parameter of Fluzoparib: t1/2 | 4 weeks
Evaluation of pharmacokinetic parameter of Fluzoparib: AUC | 4 weeks
Preliminary antitumor activity for the regimen, objective response rate(ORR) | 8 weeks
  To evaluate ORR 8 weeks after the initiation of Fluzoparib
Number of participants with adverse events. | 8 weeks
  Number of Participants with treatment related Adverse Events as Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - No.307 Hospital, Academy of Military Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality